CLINICAL TRIAL: NCT02492958
Title: A Phase 1/2a Placebo-controlled, Randomized, Double-blind, Sponsor-unblinded Trial To Evaluate The Safety, Tolerability, And Immunogenicity Of Staphylococcus Aureus 4-antigen Vaccine (sa4ag) In Japanese Adults
Brief Title: SA4Ag Safety, Tolerability, and Immunogenicity Study in Japanese Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: B3451003; 6123K1-1006 (Other: Alias Study Number)
Record Dates: First submitted 2015-05-29; First posted 2015-07-09 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Staphylococcal Infections
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SA4Ag (Experimental): Staphylococcus aureus 4-antigen vaccine
  Interventions: Biological: Staphylococcus aureus 4-antigen vaccine
- Placebo (Placebo Comparator): a lyophile match to the vaccine, consisting of excipients of SA4Ag formulation minus the active ingredients
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Staphylococcus aureus 4-antigen vaccine — a single 0.5 mL dose of investigational product into the deltoid muscle in the upper arm
  Other Names: SA4Ag
  Arms: SA4Ag
Biological: Placebo — a single 0.5 mL dose of investigational product into the deltoid muscle in the upper arm
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of a single dose of Staphylococcus aureus 4 antigen vaccine in Japanese adults aged 20 to <86 years.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese male and female adults aged 20 to <86 years,
2. Determined as healthy by the investigator (Subjects with preexisting chronic medical conditions determined to be stable may be included),
3. Must be available for the 12 month duration of the study,
4. Subjects must agree to use an acceptable method of birth control for 3 months after study vaccination (if the subject or the subject's partner are/is capable of having children).

Exclusion Criteria:

1. Any contraindication to vaccination or vaccine components, including previous anaphylactic reaction to any vaccine or vaccine-related components,
2. Unstable or serious chronic medical condition that would increase the subject's risk of participation,
3. Immune system suppression or treatment with medications that suppress the immune system,
4. Receipt of blood products or immunoglobulins within the past 12 months,
5. Any infection proven or suspected to be caused by S.aureus within the past 6 months,
6. A staff member at this site nor a relative of those site staff members, nor a sponsor's employee directly involved in the conduct of this research study,
7. Living in a nursing home, long-term care facility or other institution or requiring any types of nursing care,
8. A pregnant or a breast feeding woman.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Japan (2):
  - SOUSEIKAI Sumida Hospital (formerly Medical Co. LTA Sumida Hospital), Sumida-ku, Tokyo
  - SOUSEIKAI PS Clinic (formerly Medical Co. LTA PS Clinic), Fukuoka

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3451003&StudyName=A%20Phase%201%2F2a%20Placebo-controlled%2C%20Randomized%2C%20Double-blind%2C%20Sponsor-unblinded%20Trial%20To%20Evaluate%20The%20Safety%2C%20Tolerability%2C%20And%20Immunogenicity%20Of%20Staphylococcus%20Aureus%204-antigen%20Vaccine%20%28sa4ag%29%20In%20Japanese%20Adults

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (20 to <65 Years): Participants aged from 20 years to less than (<) 65 years, received a single dose of placebo matched to Staphylococcus aureus 4-antigen (SA4Ag) vaccine intramuscularly on Day 1. Participants were followed up to Month 12.
- SA4Ag (20 to <65 Years): Participants aged from 20 years to <65 years, received a single 0.5 milliliter (mL) dose of SA4Ag vaccine intramuscularly on Day 1. Participants were followed up to Month 12.
- Placebo (65 to <86 Years): Participants aged from 65 years to <86 years, received a single dose of placebo matched to SA4Ag vaccine intramuscularly on Day 1. Participants were followed up to Month 12.
- SA4Ag (65 to <86 Years): Participants aged from 65 years to <86 years, received a single 0.5 mL dose of SA4Ag vaccine intramuscularly on Day 1. Participants were followed up to Month 12.
Period: Overall Study
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Started | 34 | 34 | 34 | 34
Completed | 33 | 34 | 32 | 34
Not Completed | 1 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of investigational product and had safety data available after vaccination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years) | Total
Number analyzed (Participants) | 34 | 34 | 34 | 34 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 (12.2) | 0 (12.1) | 0 (4.2) | 0 (3.6) | 0
  Between 18 and 65 years | 34 | 34 | 0 | 0 | 68
  >=65 years | 0 | 0 | 34 | 34 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 21 | 13 | 68
  Male | 15 | 19 | 13 | 21 | 68

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With At Least 1 Local Reaction Within 14 Days of Vaccination
Description: Local reactions were recorded using an electronic daily diary. Local reactions included redness, swelling and pain at injection site. Redness and swelling were defined as mild (2.5 to 5.0 centimeters [cm]), moderate (5.5 to 10.0 cm) and, severe (greater than or equal to [>=] 10.5 cm). Pain at injection site was defined as mild (did not interfere with activity), moderate (interfered with activity), and severe (prevented daily activity). In this outcome measure percentage of participants with any local reaction was reported.
Time Frame: Day 1 up to Day 14
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Percentage of participants | 2.9 [0.1 to 15.3] | 20.6 [8.7 to 37.9] | 5.9 [0.7 to 19.7] | 29.4 [15.1 to 47.5]

2. Primary Outcome: Percentage of Participants With Local Reactions by Severity Within 14 Days of Vaccination
Description: Local reactions were recorded using an electronic daily diary. Local reactions included redness, swelling and pain at injection site. Redness and swelling were graded as mild (2.5 to 5.0 cm), moderate (5.5 to 10.0 cm) and, severe (>=10.5 cm). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), and severe (prevented daily activity).
Time Frame: Day 1 up to Day 14
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Percentage of participants
  Redness: Mild | 2.9 [0.1 to 15.3] | 2.9 [0.1 to 15.3] | 2.9 [0.1 to 15.3] | 5.9 [0.7 to 19.7]
  Redness: Moderate | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 5.9 [0.7 to 19.7]
  Redness: Severe | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 2.9 [0.1 to 15.3]
  Swelling: Mild | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 5.9 [0.7 to 19.7] | 0.0 [0.0 to 10.3]
  Swelling: Moderate | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 8.8 [1.9 to 23.7]
  Swelling: Severe | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3]
  Pain: Mild | 0.0 [0.0 to 10.3] | 17.6 [6.8 to 34.5] | 2.9 [0.1 to 15.3] | 14.7 [5.0 to 31.1]
  Pain: Moderate | 0.0 [0.0 to 10.3] | 2.9 [0.1 to 15.3] | 0.0 [0.0 to 10.3] | 5.9 [0.7 to 19.7]
  Pain: Severe | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3]

3. Primary Outcome: Percentage of Participants With At Least 1 Systemic Event Within 14 Days of Vaccination
Description: Systemic reactions included fever, vomiting, diarrhea, headache, fatigue, muscle and joint pain (other than at the injection site) and recorded by using an e-diary. Fever was graded as 37.5 to 38.4 degree Celsius (C), 38.5 to 38.9 degree C, 39.0 to 40.0 degree C and greater than (>) 40.0 degree C. Vomiting was graded as mild (1-2 times in 24 hours), moderate (>2 times in 24 hours) and severe (required intravenous hydration). Diarrhea was graded as mild (2-3 loose stools in 24 hours), moderate (4-5 loose stools in 24 hours) and severe (>=6 loose stools in 24 hours). Headache, fatigue, muscle pain and joint pain were graded as mild (no interference with activity), moderate (some interference with activity) and severe (significant, prevented daily activity). In this outcome measure percentage of participants with any systemic event was reported.
Time Frame: Day 1 up to Day 14
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Percentage of participants | 29.4 [15.1 to 47.5] | 29.4 [15.1 to 47.5] | 17.6 [6.8 to 34.5] | 35.3 [19.7 to 53.5]

4. Primary Outcome: Percentage of Participants With Systemic Events by Severity Within 14 Days of Vaccination
Description: Systemic reactions included fever, vomiting, diarrhea, headache, fatigue, muscle and joint pain (other than at the injection site) and recorded by using an e-diary. Fever was graded as 37.5 to 38.4 degree C, 38.5 to 38.9 degree C, 39.0 to 40.0 degree C and >40.0 degree C. Vomiting was graded as mild (1-2 times in 24 hours), moderate (>2 times in 24 hours) and severe (required intravenous hydration). Diarrhea was graded as mild (2-3 loose stools in 24 hours), moderate (4-5 loose stools in 24 hours) and severe (>=6 loose stools in 24 hours). Headache, fatigue, muscle pain and joint pain were graded as mild (no interference with activity), moderate (some interference with activity) and severe (significant, prevented daily activity).
Time Frame: Day 1 up to Day 14
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Percentage of participants
  Fever: 37.5 degree C-38.4 degree C | 0.0 [0.0 to 10.3] | 5.9 [0.7 to 19.7] | 2.9 [0.1 to 15.3] | 5.9 [0.7 to 19.7]
  Fever: 38.5 degree C-38.9 degree C | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3]
  Fever: 39.0 degree C-40.0 degree C | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3]
  Fever: >40.0 degree C | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3]
  Fatigue: Mild | 8.8 [1.9 to 23.7] | 8.8 [1.9 to 23.7] | 5.9 [0.7 to 19.7] | 11.8 [3.3 to 27.5]
  Fatigue: Moderate | 5.9 [0.7 to 19.7] | 2.9 [0.1 to 15.3] | 0.0 [0.0 to 10.3] | 5.9 [0.7 to 19.7]
  Fatigue: Severe | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3]
  Headache: Mild | 5.9 [0.7 to 19.7] | 11.8 [3.3 to 27.5] | 2.9 [0.1 to 15.3] | 5.9 [0.7 to 19.7]
  Headache: Moderate | 5.9 [0.7 to 19.7] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 2.9 [0.1 to 15.3]
  Headache: Severe | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3]
  Vomiting: Mild | 2.9 [0.1 to 15.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3]
  Vomiting: Moderate | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3]
  Vomiting: Severe | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3]
  Diarrhea: Mild | 14.7 [5.0 to 31.1] | 5.9 [0.7 to 19.7] | 0.0 [0.0 to 10.3] | 5.9 [0.7 to 19.7]
  Diarrhea: Moderate | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3]
  Diarrhea: Severe | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3]
  Muscle Pain: Mild | 0.0 [0.0 to 10.3] | 2.9 [0.1 to 15.3] | 8.8 [1.9 to 23.7] | 8.8 [1.9 to 23.7]
  Muscle Pain: Moderate | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 5.9 [0.7 to 19.7]
  Muscle Pain: Severe | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3]
  Joint Pain: Mild | 0.0 [0.0 to 10.3] | 2.9 [0.1 to 15.3] | 0.0 [0.0 to 10.3] | 5.9 [0.7 to 19.7]
  Joint Pain: Moderate | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 2.9 [0.1 to 15.3]
  Joint Pain: Severe | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 10.3]

5. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) Reported From Day 1 Up to Day 29 Visit
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AEs included both serious and non-serious AEs. Treatment-emergent AEs were events between the administration of investigational product and up to Day 29 that were absent before vaccination or that worsened relative to pre-administration state.
Time Frame: Day 1 up to Day 29
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Percentage of participants | 5.9 | 2.9 | 5.9 | 5.9

6. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAE) Reported After Day 29 Visit Through Month 12
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or deemed medically significant for any other reason. A treatment emergent AE was defined as an event that emerged during the study that was absent before administration of investigational product, or worsened relative to the pre-administration state. AEs reported during this time period included both SAEs and newly diagnosed chronic medical disorders (NDCMD). A NDCMD was defined as a disease or medical condition that was not identified prior to study start and was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: After Day 29 up to Month 12
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Percentage of participants
  AEs | 2.9 | 0.0 | 5.9 | 11.8
  SAEs | 2.9 | 0.0 | 5.9 | 8.8

7. Primary Outcome: Percentage of Participants With Hematology Abnormalities at Day 5
Description: Hematology analysis included the following parameters: hemoglobin, white blood cells, neutrophils and platelets, and scaled as Grade 1= mild; Grade 2= moderate; Grade 3= severe; or Grade 4. Hematology abnormality was defined as at least 1 grade abnormal value. Percentage of participants with abnormal values in hematology parameters are reported in this outcome measure.
Time Frame: Day 5
Population: Safety population included all participants who received at least 1 dose of investigational product and had safety data available after vaccination. Here 'number of participants analyzed (N)' signifies number of participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Percentage of participants
  Hemoglobin | 0.0 | 16.7 | 0.0 | 0.0
  White Blood Cells | 0.0 | 16.7 | 0.0 | 0.0
  Neutrophils | 0.0 | 33.3 | 0.0 | 16.7
  Platelets | 0.0 | 0.0 | 0.0 | 0.0

8. Primary Outcome: Percentage of Participants With Hematology Abnormalities at Day 15
Description: as for outcome 7
Time Frame: Day 15
Population: Safety population included all participants who received at least 1 dose of investigational product and had safety data available after vaccination. Here N signifies number of participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Percentage of participants
  Hemoglobin | 16.7 | 50.0 | 0.0 | 16.7
  White Blood Cells | 0.0 | 33.3 | 0.0 | 0.0
  Neutrophils | 0.0 | 33.3 | 0.0 | 16.7
  Platelets | 0.0 | 0.0 | 0.0 | 0.0

9. Primary Outcome: Percentage of Participants With Coagulation Abnormalities at Day 5
Description: Coagulation analysis included the following parameters: prothrombin time (PT), activated partial thromboplastin time (APTT), platelet aggregation (AGG) (with adenosine diphosphate [ADP], with arachidonic acid, and with collagen) and fibrinogen activity. PT and APTT were scaled as Grade 1= mild; Grade 2= moderate; Grade 3= severe; or Grade 4. Coagulation abnormality was defined as at least 1 grade abnormal value for PT and APTT, and deviation from local laboratory range for platelet aggregation assay and fibrinogen activity assay. Percentage of participants with abnormal values in coagulation parameters are reported in this outcome measure.
Time Frame: Day 5
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Percentage of participants
  PT | 0.0 | 0.0 | 0.0 | 0.0
  APTT | 0.0 | 0.0 | 0.0 | 0.0
  Platelet AGG: ADP | 0.0 | 0.0 | 0.0 | 0.0
  Platelet AGG: Arachidonic acid | 0.0 | 0.0 | 33.3 | 0.0
  Platelet AGG: Collagen | 0.0 | 0.0 | 0.0 | 0.0
  Fibrinogen Activity | 0.0 | 0.0 | 0.0 | 16.7

10. Primary Outcome: Percentage of Participants With Coagulation Abnormalities at Day 15
Description: Coagulation analysis included the following parameters: PT, APTT, platelet AGG with ADP, platelet AGG with arachidonic acid, platelet AGG with collagen and fibrinogen activity. PT and APTT were scaled as Grade 1= mild; Grade 2= moderate; Grade 3= severe; or Grade 4. Coagulation abnormality was defined as at least 1 grade abnormal value for PT and APTT, and deviation from local laboratory range for platelet aggregation assay and fibrinogen activity assay. Percentage of participants with abnormal values in coagulation parameters are reported in this outcome measure.
Time Frame: Day 15
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Percentage of participants
  PT | 0.0 | 0.0 | 0.0 | 0.0
  APTT | 0.0 | 0.0 | 0.0 | 0.0
  Platelet AGG: ADP | 0.0 | 0.0 | 0.0 | 0.0
  Platelet AGG: Arachidonic acid | 0.0 | 0.0 | 0.0 | 16.7
  Platelet AGG: Collagen | 0.0 | 0.0 | 0.0 | 0.0
  Fibrinogen Activity | 0.0 | 0.0 | 0.0 | 0.0

11. Primary Outcome: Percentage of Participants With Blood Chemistry Abnormalities at Day 5
Description: Blood chemistry laboratory analysis included the following parameters: alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, bilirubin, creatinine, creatine kinase and lactate dehydrogenase, and scaled as Grade 1= mild; Grade 2= moderate; Grade 3= severe; or Grade 4. Blood chemistry abnormality was defined as at least 1 grade abnormal value. Percentage of participants with abnormal values in blood chemistry laboratory parameters are reported in this outcome measure.
Time Frame: Day 5
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Percentage of participants
  Alanine Aminotransferase | 0.0 | 0.0 | 0.0 | 0.0
  Aspartate Aminotransferase | 0.0 | 0.0 | 0.0 | 0.0
  Alkaline Phosphatase | 0.0 | 0.0 | 0.0 | 16.7
  Bilirubin | 0.0 | 16.7 | 0.0 | 0.0
  Creatinine | 0.0 | 0.0 | 0.0 | 0.0
  Creatine Kinase | 0.0 | 33.3 | 0.0 | 0.0
  Lactate Dehydrogenase | 16.7 | 16.7 | 0.0 | 16.7

12. Primary Outcome: Percentage of Participants With Blood Chemistry Abnormalities at Day 15
Description: as for outcome 11
Time Frame: Day 15
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Percentage of participants
  Alanine Aminotransferase | 0.0 | 0.0 | 0.0 | 0.0
  Aspartate Aminotransferase | 0.0 | 0.0 | 0.0 | 0.0
  Alkaline Phosphatase | 0.0 | 0.0 | 0.0 | 16.7
  Bilirubin | 0.0 | 0.0 | 16.7 | 0.0
  Creatinine | 0.0 | 0.0 | 0.0 | 0.0
  Creatine Kinase | 0.0 | 0.0 | 16.7 | 0.0
  Lactate Dehydrogenase | 16.7 | 0.0 | 16.7 | 16.7

13. Primary Outcome: Percentage of Participants Achieving Predefined Antibody Response to Target Antigens at Day 29
Description: Percentage of participants achieving predefined antibody response to capsular polysaccharide serotype 5 (CP5), capsular polysaccharide serotype 8 (CP8), clumping factor A (ClfA) and manganese transporter C (MntC) at Day 29 were reported. The predefined thresholds for the target antigens were 1000 and 2000 based on opsonophagocytic activity (OPA) assay for CP5 and CP8, respectively; was 121 based on fibrinogen-binding inhibition (FBI) assay for ClfA and 512 based on competitive Luminex immunoassay (cLIA) for MntC.
Time Frame: Day 29
Population: The evaluable immunogenicity population included all participants who received investigational product to which they were randomized, had valid and determinate assay result for at least 1 antigen for primary immunogenicity analysis. Here "n" signifies the number of participants who were evaluable for specific antigens for each arm, respectively.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Percentage of participants
  CP5: number analyzed (Participants) | 31 | 34 | 32 | 34
  CP5 | 25.8 [11.9 to 44.6] | 100.0 [89.7 to 100.0] | 15.6 [5.3 to 32.8] | 100.0 [89.7 to 100.0]
  CP8 | 17.6 [6.8 to 34.5] | 100.0 [89.7 to 100.0] | 20.6 [8.7 to 37.9] | 94.1 [80.3 to 99.3]
  ClfA | 8.8 [1.9 to 23.7] | 94.1 [80.3 to 99.3] | 5.9 [0.7 to 19.7] | 88.2 [72.5 to 96.7]
  MntC | 2.9 [0.1 to 15.3] | 91.2 [76.3 to 98.1] | 8.8 [1.9 to 23.7] | 94.1 [80.3 to 99.3]

14. Secondary Outcome: Percentage of Participants Achieving Predefined Antibody Response to Target Antigens on Baseline, Day 11, 15 and Month 3
Description: Percentage of participants achieving predefined antibody response to CP5, CP8, ClfA and MntC at Baseline, Day 11, 15 and Month 3 were reported. The predefined thresholds for the target antigens were 1000 and 2000 based on OPA assay for CP5 and CP8, respectively; was 121 based on FBI assay for ClfA, 512 based on cLIA for MntC.
Time Frame: Baseline, Day 11, 15 and Month3
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Percentage of participants
  Baseline: CP5 | 20.6 [8.7 to 37.9] | 23.5 [10.7 to 41.2] | 11.8 [3.3 to 27.5] | 14.7 [5.0 to 31.1]
  Baseline: CP8: number analyzed (Participants) | 33 | 33 | 34 | 34
  Baseline: CP8 | 15.2 [5.1 to 31.9] | 33.3 [18.0 to 51.8] | 20.6 [8.7 to 37.9] | 26.5 [12.9 to 44.4]
  Baseline: ClfA | 11.8 [3.3 to 27.5] | 0.0 [0.0 to 10.3] | 2.9 [0.1 to 15.3] | 0.0 [0.0 to 10.3]
  Baseline: MntC | 2.9 [0.1 to 15.3] | 23.5 [10.7 to 41.2] | 8.8 [1.9 to 23.7] | 11.8 [3.3 to 27.5]
  Day 11: CP5: number analyzed (Participants) | 34 | 33 | 33 | 34
  Day 11: CP5 | 20.6 [8.7 to 37.9] | 100.0 [89.4 to 100.0] | 18.2 [7.0 to 35.5] | 100.0 [89.7 to 100.0]
  Day 11: CP8: number analyzed (Participants) | 33 | 34 | 34 | 34
  Day 11: CP8 | 18.2 [7.0 to 35.5] | 100.0 [89.7 to 100.0] | 20.6 [8.7 to 37.9] | 94.1 [80.3 to 99.3]
  Day 11: ClfA | 11.8 [3.3 to 27.5] | 97.1 [84.7 to 99.9] | 2.9 [0.1 to 15.3] | 82.4 [65.5 to 93.2]
  Day 11: MntC | 2.9 [0.1 to 15.3] | 94.1 [80.3 to 99.3] | 8.8 [1.9 to 23.7] | 97.1 [84.7 to 99.9]
  Day 15: CP5: number analyzed (Participants) | 33 | 34 | 33 | 34
  Day 15: CP5 | 21.2 [9.0 to 38.9] | 100.0 [89.7 to 100.0] | 9.1 [1.9 to 24.3] | 100.0 [89.7 to 100.0]
  Day 15: CP8: number analyzed (Participants) | 32 | 34 | 34 | 34
  Day 15: CP8 | 18.8 [7.2 to 36.4] | 100.0 [89.7 to 100.0] | 20.6 [8.7 to 37.9] | 97.1 [84.7 to 99.9]
  Day 15: ClfA | 11.8 [3.3 to 27.5] | 97.1 [84.7 to 99.9] | 5.9 [0.7 to 19.7] | 88.2 [72.5 to 96.7]
  Day 15: MntC | 2.9 [0.1 to 15.3] | 94.1 [80.3 to 99.3] | 17.6 [6.8 to 34.5] | 97.1 [84.7 to 99.9]
  Month 3: CP5: number analyzed (Participants) | 32 | 34 | 34 | 34
  Month 3: CP5 | 18.8 [7.2 to 36.4] | 100.0 [89.7 to 100.0] | 20.6 [8.7 to 37.9] | 100.0 [89.7 to 100.0]
  Month 3: CP8 | 20.6 [8.7 to 37.9] | 100.0 [89.7 to 100.0] | 14.7 [5.0 to 31.1] | 88.2 [72.5 to 96.7]
  Month 3: ClfA | 2.9 [0.1 to 15.3] | 88.2 [72.5 to 96.7] | 2.9 [0.1 to 15.3] | 82.4 [65.5 to 93.2]
  Month 3: MntC | 2.9 [0.1 to 15.3] | 76.5 [58.8 to 89.3] | 14.7 [5.0 to 31.1] | 82.4 [65.5 to 93.2]

15. Secondary Outcome: Antigen-specific Competitive Luminex Immunoassay (cLIA) Geometric Mean Titers (GMTs)
Description: Geometric mean titer is commonly used to assess the immunogenicity of vaccine. Antibody GMTs as measured by cLIA for ClfA and MntC and corresponding 2-sided 95 percent (%) confidence intervals (CIs) were evaluated. CIs were computed by back transforming the CIs generated for means of the titers on the log scale based on the Student t distribution.
Time Frame: Baseline, Day 11, 15, 29 and Month 3
Population: The evaluable immunogenicity population included all participants who received the investigational product to which they were randomized, had valid and determinate assay result for at least 1 antigen for the primary immunogenicity analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Titer
  Baseline: ClfA | 200.7 [177.6 to 226.8] | 218.1 [196.7 to 241.7] | 216.6 [179.7 to 261.0] | 174.0 [150.3 to 201.4]
  Baseline: MntC | 349.4 [306.8 to 398.0] | 376.8 [316.5 to 448.5] | 321.4 [270.6 to 381.7] | 334.8 [291.6 to 384.3]
  Day 11: ClfA | 190.7 [166.1 to 218.9] | 4105.2 [2389.4 to 7053.0] | 203.7 [172.2 to 241.0] | 3394.1 [2029.3 to 5676.8]
  Day 11: MntC | 358.5 [312.2 to 411.6] | 5019.6 [3207.2 to 7856.2] | 313.6 [260.9 to 377.0] | 6712.9 [4385.4 to 10275.6]
  Day 15: ClfA | 198.7 [172.2 to 229.2] | 4706.0 [2802.7 to 7902.1] | 231.9 [199.1 to 270.1] | 4571.3 [2883.1 to 7248.1]
  Day 15: MntC | 351.4 [312.2 to 395.6] | 4431.7 [2896.0 to 6781.7] | 356.0 [297.8 to 425.5] | 5710.0 [3816.9 to 8541.9]
  Day 29: ClfA | 198.4 [173.7 to 226.6] | 3815.0 [2288.8 to 6359.0] | 182.5 [149.4 to 223.1] | 3313.6 [2155.0 to 5095.3]
  Day 29: MntC | 326.9 [287.2 to 371.9] | 2920.8 [1947.4 to 4380.8] | 281.4 [235.8 to 335.7] | 3471.0 [2397.3 to 5025.5]
  Month 3: ClfA | 201.6 [177.3 to 229.2] | 2309.3 [1492.9 to 3572.3] | 224.8 [190.8 to 264.8] | 2054.8 [1348.3 to 3131.6]
  Month 3: MntC | 316.3 [275.6 to 363.0] | 1273.5 [912.1 to 1778.0] | 384.1 [329.9 to 447.2] | 1528.7 [1112.2 to 2101.1]

16. Secondary Outcome: Antigen-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs)
Description: Geometric mean titer is commonly used to assess the immunogenicity of vaccine. Antibody GMTs as measured by OPA for CP5 and CP8 and corresponding 2-sided 95 percent CIs were evaluated. CIs were computed by back transforming the CIs generated for means of the titers on the log scale based on the Student t distribution.
Time Frame: Baseline, Day 11, 15, 29 and Month 3
Population: The evaluable immunogenicity population included all participants who received the investigational product to which they were randomized, had valid and determinate assay result for at least 1 antigen for primary immunogenicity analysis. Here "n" signifies number of participants who were evaluable for specific antigens for each arm, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Titer
  Baseline: CP5 | 355.1 [227.7 to 553.8] | 301.7 [197.4 to 461.0] | 349.0 [249.2 to 488.9] | 332.9 [223.9 to 495.1]
  Baseline: CP8: number analyzed (Participants) | 33 | 33 | 34 | 34
  Baseline: CP8 | 512.9 [338.4 to 777.5] | 702.5 [407.8 to 1210.1] | 337.3 [195.7 to 581.3] | 388.6 [222.6 to 678.3]
  Day 11: CP5: number analyzed (Participants) | 34 | 33 | 33 | 34
  Day 11: CP5 | 360.6 [231.7 to 561.1] | 37617.8 [27863.0 to 50787.8] | 342.0 [231.1 to 506.2] | 31066.0 [20279.0 to 47591.1]
  Day 11: CP8: number analyzed (Participants) | 33 | 34 | 34 | 34
  Day 11: CP8 | 567.9 [372.3 to 866.3] | 27501.3 [19669.7 to 38451.2] | 351.2 [205.9 to 598.9] | 16214.6 [8218.2 to 31991.7]
  Day 15: CP5: number analyzed (Participants) | 33 | 34 | 33 | 34
  Day 15: CP5 | 354.9 [236.9 to 531.9] | 26677.0 [20149.0 to 35319.9] | 331.3 [231.2 to 474.9] | 31706.4 [21585.9 to 46571.8]
  Day 15: CP8: number analyzed (Participants) | 32 | 34 | 34 | 34
  Day 15: CP8 | 514.7 [333.8 to 793.5] | 25403.8 [18448.2 to 34981.9] | 326.6 [193.6 to 551.1] | 24039.8 [13014.0 to 44407.0]
  Day 29: CP5: number analyzed (Participants) | 31 | 34 | 32 | 34
  Day 29: CP5 | 432.6 [275.3 to 679.8] | 25026.5 [18911.3 to 33119.1] | 350.1 [241.8 to 506.9] | 29639.2 [20983.3 to 41865.7]
  Day 29: CP8 | 544.5 [362.0 to 819.1] | 23453.9 [16904.7 to 32540.3] | 336.4 [195.7 to 578.3] | 16542.0 [9489.2 to 28836.7]
  Month 3: CP5: number analyzed (Participants) | 32 | 34 | 34 | 34
  Month 3: CP5 | 410.0 [266.1 to 631.8] | 14679.2 [11032.9 to 19530.7] | 339.8 [238.9 to 483.4] | 16000.3 [11448.0 to 22362.8]
  Month 3: CP8 | 504.1 [327.4 to 776.2] | 11856.2 [8663.2 to 16226.1] | 308.5 [187.1 to 508.7] | 7881.5 [4521.6 to 13738.1]

17. Secondary Outcome: Antigen-specific Fibrinogen-binding Inhibition (FBI) Assay Geometric Mean Titers (GMTs)
Description: Geometric mean titer is commonly used to assess the immunogenicity of vaccine. Antibody GMTs as measured by FBI for ClfA and corresponding 2-sided 95 percent CIs were evaluated. CIs were computed by back transforming the CIs generated for means of the titers on the log scale based on the Student t distribution.
Time Frame: Baseline, Day 11, 15, 29 and Month 3
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Titer
  Baseline | 67.2 [60.5 to 74.7] | 60.5 [NA to NA] — CI was not estimated due to the lack of variability of GMT. | 63.3 [57.7 to 69.4] | 60.5 [NA to NA] — CI was not estimated due to the lack of variability of GMT.
  Day 11 | 68.4 [59.7 to 78.3] | 755.5 [468.1 to 1219.2] | 63.3 [57.7 to 69.4] | 620.1 [367.8 to 1045.6]
  Day 15 | 69.9 [60.2 to 81.2] | 868.5 [544.1 to 1386.3] | 64.6 [58.7 to 71.1] | 706.8 [421.2 to 1185.9]
  Day 29 | 68.1 [59.1 to 78.5] | 748.4 [473.0 to 1184.4] | 65.2 [58.6 to 72.5] | 620.7 [396.5 to 971.8]
  Month 3 | 64.0 [57.1 to 71.8] | 474.5 [309.7 to 726.9] | 63.1 [57.9 to 68.8] | 384.8 [256.1 to 578.3]

18. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for Staphylococcus Aureus Antigen-specific cLIA Titers From Baseline to Day 11, 15, 29 and Month 3
Description: GMFRs of anti-Staphylococcus aureus cLIA for ClfA and MntC were computed. CIs which are reported below were computed by back transforming the CIs generated for the mean fold rise on the log scale based on the Student t distribution. GMFRs were computed as the fold rise in titer value at specified time point compared to baseline.
Time Frame: Baseline, Day 11, 15, 29 and Month 3
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Fold rise
  Day 11: ClfA | 1.0 [0.9 to 1.0] | 18.8 [11.0 to 32.1] | 0.9 [0.9 to 1.0] | 19.5 [12.0 to 31.8]
  Day 11: MntC | 1.0 [0.9 to 1.1] | 13.3 [9.0 to 19.8] | 1.0 [0.9 to 1.1] | 20.1 [13.2 to 30.5]
  Day 15: ClfA | 1.0 [0.9 to 1.1] | 21.6 [13.0 to 35.7] | 1.1 [1.0 to 1.2] | 26.3 [17.0 to 40.5]
  Day 15: MntC | 1.0 [0.9 to 1.1] | 11.8 [8.1 to 17.1] | 1.1 [1.0 to 1.3] | 17.1 [11.5 to 25.3]
  Day 29: ClfA | 1.0 [0.9 to 1.1] | 17.5 [10.7 to 28.7] | 0.8 [0.8 to 0.9] | 19.0 [12.8 to 28.4]
  Day 29: MntC | 0.9 [0.8 to 1.1] | 7.8 [5.5 to 10.9] | 0.9 [0.8 to 1.0] | 10.4 [7.3 to 14.7]
  Month 3: ClfA | 1.0 [0.9 to 1.1] | 10.6 [7.0 to 16.1] | 1.0 [1.0 to 1.1] | 11.8 [8.0 to 17.5]
  Month 3: MntC | 0.9 [0.8 to 1.0] | 3.4 [2.6 to 4.4] | 1.2 [1.1 to 1.4] | 4.6 [3.4 to 6.1]

19. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for Staphylococcus Aureus Antigen-specific OPA Titers From Baseline to Day 11, 15, 29 and Month 3
Description: GMFRs of anti-Staphylococcus aureus OPA for CP5 and CP8 were computed. CIs which are reported below were computed by back transforming the CIs generated for the mean fold rise on the log scale based on the Student t distribution. GMFRs were computed as the fold rise in titer value at specified time point compared to baseline.
Time Frame: Baseline, Day 11, 15, 29 and Month 3
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Fold rise
  Day 11: CP5: number analyzed (Participants) | 34 | 33 | 33 | 34
  Day 11: CP5 | 1.0 [0.8 to 1.2] | 125.0 [78.5 to 198.9] | 0.9 [0.8 to 1.0] | 93.3 [56.7 to 153.5]
  Day 11: CP8: number analyzed (Participants) | 32 | 33 | 34 | 34
  Day 11: CP8 | 1.1 [1.0 to 1.3] | 38.7 [21.0 to 71.3] | 1.0 [0.9 to 1.1] | 41.7 [20.6 to 84.6]
  Day 15: CP5: number analyzed (Participants) | 33 | 34 | 33 | 34
  Day 15: CP5 | 1.0 [0.9 to 1.2] | 88.4 [59.4 to 131.6] | 0.9 [0.8 to 1.0] | 95.2 [61.5 to 147.5]
  Day 15: CP8: number analyzed (Participants) | 31 | 33 | 34 | 34
  Day 15: CP8 | 1.0 [0.9 to 1.1] | 35.2 [19.1 to 64.8] | 1.0 [0.9 to 1.0] | 61.9 [30.8 to 124.4]
  Day 29: CP5: number analyzed (Participants) | 31 | 34 | 32 | 34
  Day 29: CP5 | 1.1 [1.0 to 1.2] | 83.0 [54.2 to 126.9] | 0.9 [0.8 to 1.1] | 89.0 [58.6 to 135.2]
  Day 29: CP8: number analyzed (Participants) | 33 | 33 | 34 | 34
  Day 29: CP8 | 1.1 [1.0 to 1.2] | 32.2 [17.4 to 59.5] | 1.0 [1.0 to 1.0] | 42.6 [22.6 to 80.4]
  Month 3: CP5: number analyzed (Participants) | 32 | 34 | 34 | 34
  Month 3: CP5 | 1.1 [1.0 to 1.3] | 48.7 [34.2 to 69.2] | 1.0 [0.9 to 1.1] | 48.1 [32.1 to 71.9]
  Month 3: CP8: number analyzed (Participants) | 33 | 33 | 34 | 34
  Month 3: CP8 | 1.0 [0.9 to 1.2] | 16.2 [9.6 to 27.6] | 0.9 [0.8 to 1.0] | 20.3 [11.5 to 35.8]

20. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for Staphylococcus Aureus Antigen-specific FBI Titers From Baseline to Day 11, 15, 29 and Month 3
Description: GMFR of anti-Staphylococcus aureus FBI for ClfA was computed. CIs which are reported below were computed by back transforming the CIs generated for the mean fold rise on the log scale based on the Student t distribution. GMFRs were computed as the fold rise in titer value at specified time point compared to baseline.
Time Frame: Baseline, Day 11, 15, 29 and Month 3
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Fold rise
  Day 11 | 1.0 [0.9 to 1.1] | 12.5 [7.7 to 20.2] | 1.0 [NA to NA] — CI was not estimated due to the lack of variability of GMFR. | 10.3 [6.1 to 17.3]
  Day 15 | 1.0 [0.9 to 1.2] | 14.4 [9.0 to 22.9] | 1.0 [1.0 to 1.1] | 11.7 [7.0 to 19.6]
  Day 29 | 1.0 [0.9 to 1.1] | 12.4 [7.8 to 19.6] | 1.0 [1.0 to 1.1] | 10.3 [6.6 to 16.1]
  Month 3 | 1.0 [0.9 to 1.0] | 7.8 [5.1 to 12.0] | 1.0 [1.0 to 1.0] | 6.4 [4.2 to 9.6]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Placebo (20 to <65 Years) | SA4Ag (20 to <65 Years) | Placebo (65 to <86 Years) | SA4Ag (65 to <86 Years)
Serious Adverse Events (participants affected / at risk) | 1/34 | 0/34 | 2/34 | 3/34
Other Adverse Events (participants affected / at risk) | 11/34 | 13/34 | 8/34 | 17/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (20 to <65 Years) (N=34) | SA4Ag (20 to <65 Years) (N=34) | Placebo (65 to <86 Years) (N=34) | SA4Ag (65 to <86 Years) (N=34)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hyalosis asteroid (Eye disorders) | 0 | 0 | 0 | 1
Macular fibrosis (Eye disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Carotid artery aneurysm (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0/15 | 0/19 | 0/13 | 1/21 — This event was gender specific.
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (20 to <65 Years) (N=34) | SA4Ag (20 to <65 Years) (N=34) | Placebo (65 to <86 Years) (N=34) | SA4Ag (65 to <86 Years) (N=34)
Diarrhea (Gastrointestinal disorders) | 5 | 2 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 5 | 4 | 2 | 6
Injection site erythema (General disorders) | 1 | 1 | 1 | 5
Injection site pain (General disorders) | 0 | 7 | 1 | 7
Injection site pain (General disorders) | 0 | 0 | 0 | 1
Injection site swelling (General disorders) | 0 | 0 | 2 | 3
Pyrexia (General disorders) | 0 | 2 | 1 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 5
Headache (Nervous system disorders) | 4 | 4 | 1 | 3
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/15 | 0/19 | 0/13 | 1/21 — This event was gender specific.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.